CLINICAL TRIAL: NCT01548547
Title: Patient Outcomes in Simulation Education (POISE) Intravenous (IV) and Lumbar Puncture (LP) Multi-institution Protocol
Acronym: POISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAE0924
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Infant Lumbar Puncture
Keywords: intravenous line; simulation education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LP mastery learning group (Experimental)
  Interventions: Other: Simulation-based mastery learning
- IV mastery learning group (Active Comparator)
  Interventions: Other: Simulation-based mastery learning

INTERVENTIONS:
Other: Simulation-based mastery learning — Hands-on coached deliberate practice on a simulator. Training until mastery achieved.

SUMMARY:
This study aims to compare the clinical efficacy of multimedia audiovisual training to hands on "practice till perfect" training for pediatric and emergency medicine residents' procedural skills. This initial study will explore the success rates on infant lumbar puncture and child intravenous access skills in post-graduate year one pediatric residents.

ELIGIBILITY:
Inclusion Criteria:

Pediatric interns at POISE network hospitals

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Rate of clinical success with lumbar puncture (LP) procedures | Up to one year
  Online performance form
Rate of clinical success with intravenous (IV) procedures | Up to one year
  Online performance form

CONTACTS AND LOCATIONS:
Overall Officials: David Kessler, MD, MSc, Principal Investigator — Columbia University; Martin Pusic, MD, PhD, Study Director — Columbia University
Locations (1):
- Columbia University, New York, New York, United States